CLINICAL TRIAL: NCT00269373
Title: PET-CT Scan as a Diagnostic Method in Unknown Primary Tumors
Brief Title: Positron Emission Tomography - Computed Tomography (PET-CT) Scan as a Diagnostic Method in Unknown Primary Tumors
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Gedske Daugaard, Associate professor, Rigshospitalet, Denmark
Other Study IDs: 01 283694
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Unknown Primary Tumor
Keywords: Unknown primary tumor; PET-CT
MeSH Terms: conditions — Neoplasms, Unknown Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: PET-CT — no drugs included

SUMMARY:
Is PET-CT scan better than PET or CT alone in diagnosing primary tumours in patients with unknown primary tumors? Can information obtained with PET-CT replace other clinical and radiological investigations? Is PET/CT cost-effective?

DETAILED DESCRIPTION:
Patients who fulfill the international definition of unknown primary tumors can be included, except:

* Young men (<55 years) with growing mid-line tumors where a germ cell tumor could be expected will not be included.
* Patients with lymph-node metastases with squamous cell carcinoma in the head and neck region will not be included.
* Women with adenocarcinoma in lymph nodes in the axilla will not be included.

ELIGIBILITY:
Inclusion Criteria:

* Unknown primary tumors

Exclusion Criteria:

* Young men (<55 years) with growing mid-line tumors where a germ cell tumor could be expected will not be included.
* Patients with lymph-node metastases with squamous cell carcinoma in the head and neck region will not be included
* Women with adenocarcinoma in lymph nodes in the axilla will not be included

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unknown tumors
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2005-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gedske Daugaard, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark